CLINICAL TRIAL: NCT05550857
Title: Comparative Effect of Myofacial Release With and Without Eccentric Resistance on Pain, Range of Motion and Functional Disability in Patients With Achilles Tendonitis
Brief Title: Effect of Myofacial Release vs. Eccentric Resistance on Pain, ROM and Functional Disability on Achilles Tendonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha Jamil, Dr. Ayesha Jamil, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Muhammad sufyan karamat
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Achilles Tendonitis
Keywords: Physiotherapy ,; Myofascial release; Eccentric Resistance; Achilles tendonitis; Pain; Range of motion; Functional Disability
MeSH Terms: conditions — Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release (Active Comparator): Group A:
  This group will receive routine physiotherapy with myofascial release. This protocol will be given for 3 alternative days per week. Each session will be of 45 minutes. Data will be collected at baseline, at 2nd week and at 4th week.
  Interventions: Other: myofascial release
- eccentric resistance exercise (Experimental): Group B:
  This group will receive routine physiotherapy and myofascial release with eccentric resistance exercise . This protocol will be given for 3 alternative days per week. Each session will be of 60 minutes. Data will be collected at baseline, at 2nd week and at 4th week.
  Interventions: Other: eccentric resistance exercise

INTERVENTIONS:
Other: eccentric resistance exercise — The subject will lying prone on a treatment table. One end of eccentric resistance band will tie around the mid of the foot of indvidual, the other end of the resistance band will be attach to the table and the band is adjusted so that it will tight and there will be no slack present in it. It will provide a smooth eccentric resistance throughout the dorsiflexion range
  Arms: eccentric resistance exercise
Other: myofascial release — The subject will lye prone on a treatment table. Deep longitudinal massage with the help of both thumbs reinforcing eachother will be given on the subject's calf muscles.
  Arms: Myofascial release

SUMMARY:
Achilles tendinitis is a common condition that cause pain along back of leg near the heal. It is an overuse injury of the Achilles tendon, the band of tissue that connect calf muscles at the back of the lower leg to heel bone. There are number of treatment approaches to relieve pain in Achilles tendonitis . Insufficient literature has discuss the combine effect of myofascial release with eccentric resistance. So the aim of the study is to compare the effect of myofascial release with eccentric resistance and without eccentric resistance on pain , range of motion and functional disability in patient with Achilles tendinitis

DETAILED DESCRIPTION:
Tendonitis refers to inflammation of a tendon in response to injury or disease. It causes pain, irritation, and swelling, especially following periods of activity. Achilles tendinitis (AT) is a prevalent condition across the lifespan in both active and sedentary people, and can occur in the mid tendon, tendon insertion to the calcaneus and peritendon.

Achilles tendinitis is caused by overuse of the ankle and is closely related to an individuals activity level. In the adult population (21-60 yrs old), the incidence rate is 2.35 persons per 1000. It has been reported in approximately 7%-9% of professional athletes and 6%-18% of regular runners.

People with Achilles tendinitis typically report symptoms of pain and stiffness upon weight bearing after prolonged rest and at the start of physical activity, which reduces as the activity continues . These symptoms lead to impaired performance. In more severe cases, pain and disability can be persistent with functional activities such as walking.

Physical therapists have used different methods to maintain and also to increase joint motion, and prevent deformity and dysfunction resulting from the muscle shortening. The intension of the physical therapist is to lengthen the musculo-tendinous unit, supporting connective tissue and increase the range of motion.

Soft tissue treatments are widely used for AT, but strong scientific evidence to support those treatments is lacking. The literature provides some evidence that heavy pressure and deep massage might have some positive effect on chronic tendonitis by promoting healing.

Eccentric training can be effective in the rehabilitation of patients with Achilles tendonitis. The mechanism behind these results is not clear. However, there is evidence that tendons are able to respond to repeated forces by altering their structure and composition, and, thus, their mechanical properties change

ELIGIBILITY:
Inclusion Criteria:

* Both male and female.
* Age limit 25-50 year.
* Diagnosed patients by orthopedic surgeon.
* Achilles tendon symptoms (pain) present in one limb for a minimum of two months.
* Report having pain rated at least 3 out of 10 on a numerical rating scale (NRS-11).
* Be able to walk household distances (more than 50 m) without the aid of a walker, crutches or can

Exclusion Criteria:

* History of Pregnanc.
* Having history of rheumatoid arthritis or generalized polyarthritis.
* Pervious history of Achilles tendon rupture or surgery i.e arthrodesis , club foot surgery
* History of hind foot fracture, or leg-length discrepancy of more than one-half inch.
* Taken any manual therapy in last 3 month.
* Contraindication to myofacial releas i.e skin burn or disease

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
pain intensity | change in pain intensity score will be measured at baseline , at 2nd week , at 4th week
  pain intensity will be measured by Numeric Pain Rating Scale
Range of motion | Change in range of motion score will be measured at baseline , at 2nd week , at 4th week
  Range of motion will be measured by goniometer
Functional disability | change in Function disability score will be measured at baseline, at 2nd week , at 4th week
  Functional disability will be measured by ankle foot disability index

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Immediately after publication
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending on 36th month